CLINICAL TRIAL: NCT03313986
Title: Outcomes of Surgical Correction of Penile Curvature in Adult
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Elgendy, Principal Investigator, Assiut University
Other Study IDs: Adult penile curvature
Record Dates: First submitted 2017-10-09; First posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Complication of Surgical Procedure
Keywords: penile curvature; Peyronie's disease; Nesbit
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Penile curvature in adults is divided into two main categories the first is congenital penile curvature with orthotopic meatus and the other is acquired curvature which its common causes are Peyronie's disease (PD) and previous penile surgery as for hypospadias repair.The congenital penile curvatures (CPC) which not associated with urethral malformation is a relatively uncommon condition that may present in late adolescent or early adult life. The incidence is estimated to be 0.6 % but the incidence of clinically significant CPC is much lower, as the degree of curvature and sexual dysfunction varies widely Penile curvature may lead to inability for sexual intercourse. These cases require treatment. Acquired penile curvature its most common cause is Peyronie's disease. Peyronie's disease is a fibrotic disorder of the tunica albuginea of the corpora cavernosa that is clinically defined by the presence of a palpable, inelastic tunical plaque. PD is relatively common and affects up to 20.3% of adult men to some degree.

Surgery is gold-standard for treatment of curvature in stable PD. Surgical therapy is subdivided into three main procedures: (1) plication techniques (Penile shortening procedures), (2) grafting procedures with partial plaque excision or incision followed by defect closure with various grafts, and (3) correction of deviation with simultaneous penile prosthesis implantation in patients with ED not responding to medical therapy.

In this study results of different surgical techniques in management of penile curvature will be compared.

DETAILED DESCRIPTION:
The type of surgery will be chosen according to the degree of curvature and penile length after meticulous preoperative assessment.

Preoperative evaluation

* A thorough history will be taken, with special stress on:
* Sexual history, including concomitant ED and baseline erectile function as assessed using validated questionnaires such as the International Index of Erectile Function (IIEF).
* Penile curvature ;( direction, degree, interfere with intercourse (hand assisted or not), presence of pain, home (self) photograph during erection).
* Co-morbidities like vascular disease, diabetes mellitus, and cardiac disease.
* Special habits like tobacco use and drug intake.
* History of penile trauma.
* History of previous penile surgery.

  • Physical examination including
* Measurement of stretched penile length, girth measurement, and penile sensation to touch.
* Direction and degree of penile curvature will be measured using the protractor through examination of the pharmacologically erect penis by office test using intracavernosal PGE1 (20 mg) and photograph taken during erection in the outpatient clinic.
* In cases of PD, the size, number, and position of the plaques will be assessed. • Routine evaluation for fitness before surgery. Operative techniques All surgeries will be performed under anaesthesia starting by a circumfericial degloving incision. After lateral dissection and mobilization of the neurovascular bundle, an artificial erection will be performed to assess the degree of deformity and the point of maximum curvature.

Plication On convex side of the shaft, Allis clamps are used on the greater curvature to estimate the number and length of tissue needed for plications, nonabsorbable stitches are placed into the tunica albuginea in pairs and adjusted as needed to achieve optimal straightening. The artificial erection is then released and sutures tied.

Nesbit Technique On the convex side of the shaft, excision of horizontal ellipses of the tunica albuginea on the greater curvature (with approximately 1 mm for each 10º of curvature), Allis clamps are then applied until the desired straightening is achieved. These ellipses are excised and closed transversely in a stepwise fashion until curvature is completely corrected.

Modified Nesbit Technique On the convex side of the shaft consisted of a longitudinal incision in the tunica with transverse closure (Heineke- Mikulicz principle), The length of the incision is limited to about 1 cm to prevent excessive indentation of the penis.

Length-Preserving Techniques (Grafting Technique) On the concave border of the penile shaft tunica lengthening procedures involve incising or excising the plaque, and adding graft material to cover the defect, Excision can be avoided if the surgeon is able to perform relaxing incisions on the plaque with added grafting material. The graft (usually 20% larger than the defect) is then sutured to the tunica albuginea with separate running suture, The types of graft used are autologous buccal mucosa or dermal graft.

The patients will return to outpatient clinic after discharge by 1 month and 3 months to evaluate for the postoperative results and complications.

Statistical analysis The statistical analysis will be done using SPSS 21.0 (statistical package for the social sciences).

Ethical considerations Informed written consent will be obtained from all patients after explanation of the operative details and possible postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* penile curvature more than 30degree.

Exclusion Criteria:

* Age: less than 18 years.
* Non-orthotopic meatus
* Patients with ED.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with penile curvature with failure of conservative/medical treatment (nonsurgical treatment) and patient's preference for definite results According to exclusion and inclusion criteria Attending Assiut andrology outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Correcting the curvature. | 3 months postoperative
  Measure of any residual curvature present by using the protractor.
Preserving erectile function and hardness. | 4 months
  to show any affection of erectile function by using Interarnational index of Erectile dysfunction questionnaire.
Preserving penile length. | 3 months
  to measure penile length postoperative and compare to the preoperative length
Penile sensation. | 3 months
  To show any affection of penile sensation postoperative

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Makovey I, Higuchi TT, Montague DK, Angermeier KW, Wood HM. Congenital penile curvature: update and management. Curr Urol Rep. 2012 Aug;13(4):290-7. doi: 10.1007/s11934-012-0257-x. PMID 22688922
- [Result] Devine CJ Jr, Horton CE. Chordee without hypospadias. J Urol. 1973 Aug;110(2):264-71. doi: 10.1016/s0022-5347(17)60183-6. No abstract available. PMID 4722625
- [Result] Kramer SA, Aydin G, Kelalis PP. Chordee without hypospadias in children. J Urol. 1982 Sep;128(3):559-61. doi: 10.1016/s0022-5347(17)53045-1. PMID 7120563
- [Result] Donnahoo KK, Cain MP, Pope JC, Casale AJ, Keating MA, Adams MC, Rink RC. Etiology, management and surgical complications of congenital chordee without hypospadias. J Urol. 1998 Sep;160(3 Pt 2):1120-2. doi: 10.1097/00005392-199809020-00041. PMID 9719289
- [Result] Bar Yosef Y, Binyamini J, Matzkin H, Ben-Chaim J. Midline dorsal plication technique for penile curvature repair. J Urol. 2004 Oct;172(4 Pt 1):1368-9. doi: 10.1097/01.ju.0000138341.68365.b6. PMID 15371846
- [Result] Nehra A, Alterowitz R, Culkin DJ, Faraday MM, Hakim LS, Heidelbaugh JJ, Khera M, Kirkby E, McVary KT, Miner MM, Nelson CJ, Sadeghi-Nejad H, Seftel AD, Shindel AW, Burnett AL; American Urological Association Education and Research, Inc.,. Peyronie's Disease: AUA Guideline. J Urol. 2015 Sep;194(3):745-53. doi: 10.1016/j.juro.2015.05.098. Epub 2015 Jun 9. PMID 26066402